CLINICAL TRIAL: NCT05900375
Title: Pilot-testing of a Decision Aid for Parents of Infants With Ureteropelvic Junction Obstruction (UPJO)
Brief Title: Decision Aid for Parents of Infants With UPJO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0037
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Ureteropelvic Junction Obstruction; Ureteropelvic Junction; Obstruction, Congenital
Keywords: shared decision making; pragmatic trial; congenital kidney anomaly
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Receipt of PtDA (Experimental): Parents in the intervention arm will receive a paper decision aid prior to meeting with their health care professional about their child's treatment options for UPJO.
  Interventions: Behavioral: Parent Decision Aid
- Control - Usual Care (No Intervention): Parents in the control arm will not receive a paper decision aid and instead will just receive usual care about their child's treatment options for UPJO.

INTERVENTIONS:
Behavioral: Parent Decision Aid — A paper parent decision aid in color will be provided to all patients at the time of their appointment and will aid in discussion with health care professionals.
  Arms: Intervention Arm - Receipt of PtDA

SUMMARY:
Ureteropelvic junction obstruction (UPJO) is the most common etiology of high-grade hydronephrosis, affecting approximately 4,000-10,000 infants annually in the U.S. The goal of surgical treatment of UPJO is to minimize the risk of kidney damage associated with obstruction, which may occur in 30-60% of infants with high-grade hydronephrosis.1-However, the benefit of early surgery compared to observation and potential later surgery to preserve kidney function has not been well-defined. Consequently, surgeons differ on whether to initially treat with surgery or observation, with surgical rates in the first year of life varying from 15-50% across surgical practices. These variations are important to understand, as the decision for early surgery is not without risk. Prior studies suggest that infants treated surgically are at higher risk for readmission and reoperation. Early surgery also raises concerns about neurodevelopmental effects of anesthetic exposure.

To address this gap, the purpose of this pilot test is to develop a patient decision aid (PtDA) tool and pilot test its effect on parental understanding and engagement in the decision-making process at Children's Hospital Colorado. The proposed pilot is a necessary first step in preparation for a future multicenter hybrid effectiveness-implementation trial. This work will also be used to support future studies evaluating the impact of a PtDA on surgical variations and treatment outcomes in patients with UPJO and other complex congenital urologic anomalies.

ELIGIBILITY:
Inclusion Criteria (all of following are needed):

* parents (age 18-89 years) of children age 30 days - 2 years
* child is presenting for consultation for SFU grade 3-4 Hydronephrosis at Children's Hospital Colorado
* parents/child presenting at Urology appointment where a MAG 3 is performed or has recently been performed.

Exclusion Criteria:

* does not meet age parameters
* does not have a child with a UPJO

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the SDM-Q9 scores between arms | through study completion, an average of 1 year
  The primary outcome will be differences in scores between the 9-item Shared Decision Making Questionnaire (SDM-Q9) survey scores between intervention and control arms. The SDM-Q9 is a validated survey instrument measuring patient understanding and engagement in the decision making process. The scale for each question is 1-5 and higher scores mean better parent involvment and understanding.

SECONDARY OUTCOMES:
Assess differences in treatment decisions | through study completion, an average of 1 year
  The surgical rates of each patient will be assessed in each arm. Demographic variables will be controlled for especially race, ethnicity, socioeconomic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Vemulakonda, MD, JD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Since the population affected is a small vulnerable population it is not ideal to share individual level data. Data sharing is possible if in aggregate form. Guides that are developed will be shared after publication.